CLINICAL TRIAL: NCT01251588
Title: An Extension Protocol for Participants of Genzyme-Sponsored Prospective, Randomized, Open-Label, Parallel-Group, Multicenter Study of MACI® for the Treatment of Symptomatic Articular Cartilage Defects of the Femoral Condyle Including the Trochlea
Brief Title: Extension Study for Participants of MACI00206 Study of MACI® for the Treatment of Symptomatic Articular Cartilage Defects of the Knee
Acronym: Extension
Status: Completed | Type: Observational
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MACI00809; 2009-016970-33 (EudraCT Number)
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Articular Cartilage Defects
Keywords: Cartilage legions; Symptomatic focal cartilage defects; Microfracture; MACI; Autologous chondrocyte
MeSH Terms: conditions — Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MACI: autologous cultured chondrocytes on porcine collagen membrane implant received in previous MACI00206 study
  Interventions: Biological: autologous cultured chondrocytes on porcine collagen membrane
- Microfracture: Microfracture treatment received in previous MACI00206 study
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Biological: autologous cultured chondrocytes on porcine collagen membrane — Implantation received in the previous MACI00206 study
  Other Names: MACI; matrix applied characterized autologous cultured chondrocytes
  Groups: MACI
Procedure: Microfracture — Arthroscopic Microfracture treatment received in the previous MACI00206 study
  Groups: Microfracture

SUMMARY:
To examine the 5-year efficacy and safety of MACI implant, compared with arthroscopic microfracture, in participants who received study treatment in the SUMMIT study for treatment of symptomatic articular cartilage defects of the knee.

DETAILED DESCRIPTION:
This study was an open-label, multicenter extension to the SUMMIT study designed to examine the 5-year efficacy and safety of MACI compared to arthroscopic microfracture in the treatment of articular cartilage defects of the knee in participants who received study treatment in the SUMMIT study. Follow-up to 2 years post-study treatment was completed as part of the SUMMIT study. Follow-up from 3 to 5 years post-study treatment in SUMMIT was completed in this extension study.

All 144 participants who received study treatment in the SUMMIT study were eligible for enrollment into this extension study. Participants had until the end of the visit window for the last visit of this extension study (ie, Week 260 + 6 weeks) to consent to enter this extension study.

Efficacy and safety assessments were performed at scheduled visits 3, 4, and 5 years following treatment in SUMMIT (ie, at Weeks 156, 208, and 260 postarthrotomy for patients treated with MACI implant or at Weeks 156, 208, and 260 postarthroscopy for patients treated with microfracture).

ELIGIBILITY:
Randomized and received study treatment (MACI or microfracture) in the SUMMIT study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Randomized and received study treatment (MACI or microfracture) in the SUMMIT study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (14):
- Czechia (2):
  - Urazova nemocnice v Brne, Brno
  - University Hospital Na Bulovce- Department of Orthopaedic Surgery Postgraduate Medical Institute, Prague
- France (3):
  - Polyclinique Saint-Roch, Montpellier
  - Clinique Maussins-Nollet, Paris
  - Hôpital d'instruction des Armées Robert Picqué, Villenave-d'Ornon
- Netherlands (3):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Elisabeth Ziekenhuis, Tilburg
  - University Medical Centre of Utrecht, Department of Orthopaedics, Utrecht
- St Olavs Hospital, Trondheim, Norway
- Poland (3):
  - Orthopaedic & Traumatology of Motor Organs, Independent Public Clinic Hospital, Bydgoszcz
  - Regional Centre of Knee Surgery & Arthroscopy, Regional Hospital of Traumatologic Surgery, Piekary Śląskie
  - Lekmed Medical Center, Warszewo
- Kungsbacka Närsjukhus, Kungsbacka, Sweden
- University of Oxford, Nuffield Dept. of Orthopaedic Surgery, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MACI: autologous cultured chondrocytes on porcine collagen membrane: Implantation
- Microfracture: Microfracture: Arthroscopic Microfracture
Period: Overall Study
Arm/Group | MACI | Microfracture
Started | 65 | 63
Completed | 65 | 59
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Population: The patients who did not elect to participate in the Extension study differed in their degree of response in SUMMIT relative to those who elected to participate in the Extension (ie, loss of higher-responding MACI patients and lower-responding microfracture patients).
Groups:
- Total: Total of all reporting groups
Arm/Group | MACI | Microfracture | Total
Number analyzed (Participants) | 65 | 63 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at the time of MACI or microfracture treatment
  years | 34.4 (8.94) | 32.7 (8.80) | 33.6 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 40 | 42 | 82
Region of Enrollment [Number; unit: participants]
  Czech Republic | 9 | 7 | 16
  Netherlands | 28 | 30 | 58
  Sweden | 1 | 1 | 2
  Norway | 3 | 3 | 6
  Poland | 13 | 12 | 25
  United Kingdom | 3 | 3 | 6
  France | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From MACI00206 Baseline for the Participant's Knee Injury and Osteoarthritis Outcome (KOOS) Pain and Function (Sports and Recreational Activities) Scores.
Description: The KOOS is a validated knee-specific instrument developed to assess the patients' opinion of their knee and associated problems. KOOS consists of 5 subscales: Pain, Function in sports and recreational activities, other Symptoms, Function in activities of daily living (ADL), and knee related Quality of life (QOL). A 5-point Likert scale was used to record the response to each item ranging from 0 (no problems) to 4 (extreme problems). Within each subscale, items were added up and normalized to a value between 0 (extreme problems) and 100 (no problems). Subscales are not combined to calculate a total score.
Time Frame: MACI00206 Baseline to Week 156
Population: The analysis population (n=128) consists of a subpopulation of participants enrolled in the SUMMIT study (n=144). 65 of 65 MACI treated patients and 57 of 63 microfracture-treated patients completed the KOOS at Week 156.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 57
units on a scale
  Change from Baseline in KOOS Pain | 42.14 [-36.1 to 83.3] | 35.77 [-2.8 to 83.3]
  Change from Baseline in KOOS Function | 45.63 [-20.0 to 95] | 36.95 [-23.8 to 100]

2. Secondary Outcome: Change From MACI00206 Baseline for the Participant's KOOS Pain and Function (Sports and Recreational Activities) Scores
Description: as for outcome 1
Time Frame: MACI00206 Baseline and Week 260
Population: Analysis population includes all participants who completed each KOOS subscale at Week 260.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 59
units on a scale
  Change from Baseline in KOOS Pain | 45.17 [0 to 83.3] | 38.42 [-11.1 to 88.9]
  Change from Baseline in KOOS Function: number analyzed (Participants) | 64 | 59
  Change from Baseline in KOOS Function | 47.17 [-10.0 to 95.0] | 37.56 [-20.0 to 100]

3. Secondary Outcome: Magnetic Resonance Imaging (MRI) Assessments of Degree of Defect Fill
Description: MRI was assessed by the independent blinded evaluators by means of consensus. The number of participants with a degree of defect fill of >50% is reported.
Time Frame: Week 260
Population: all participants with an MRI at Week 260
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 55
Participants | 44 | 39

4. Secondary Outcome: Proportion of Patients Who Achieve at Least a 10-point Improvement From MACI00206 Baseline in KOOS Pain and Function (Sports and Recreational Activities) Scores
Description: A responder is defined as a participant with at least a 10-point improvement in both the KOOS Pain and Function (Sports and Recreational activities) scores from MACI00206 Baseline scores.
Time Frame: Up to week 260
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 63
Participants | 51 | 46

5. Secondary Outcome: The Proportion of Patients in Each Treatment Group Assessed as Treatment Failures
Description: Patients were considered as a treatment failure if all of the following 5 criteria were met:
  1. Patient's global assessment of their knee joint compared to Baseline was the same or worse
  2. Physician's global assessment of the patient's knee joint compared to Baseline was the same, worse, or significantly worse.
  3. Percent improvement from Baseline in KOOS Pain score was less than 10%.
  4. Physician diagnostic evaluation of failure excluded etiologies (eg, meniscal tear) other than failed treatment of the index lesion.
  5. The physician decided that surgical re-treatment of the index lesion(s) was required that involved either extensive debridement for lesion expansion, violation of the subchondral bone, or ACI.
Time Frame: Years 2 through 5 post treatment (MACI or microfracture)
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 63
Participants | 1 | 1

6. Secondary Outcome: Average Time to Treatment Failure
Description: ANALYSIS NOT DONE: The planned analyses concerning time to treatment failure were not conducted due to the small number of per protocol treatment failure cases. The number of per protocol treatment failures in each treatment group are reported here.
  Patients were considered as a treatment failure if all of the following 5 criteria were met:
  1. Patient's global assessment of their knee joint compared to Baseline was the same or worse
  2. Physician's global assessment of the patient's knee joint compared to Baseline was the same, worse, or significantly worse.
  3. Percent improvement from Baseline in KOOS Pain score was less than 10%.
  4. Physician diagnostic evaluation of failure excluded etiologies (eg, meniscal tear) other than failed treatment of the index lesion.
  5. The physician decided that surgical re-treatment of the index lesion(s) was required that involved either extensive debridement for lesion expansion, violation of the subchondral bone, or ACI.
Time Frame: Up to 260 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 63
Participants | 1 | 1

7. Secondary Outcome: Change From MACI00206 Baseline in the Remaining 3 Subscales (Activities of Daily Living, Quality of Life, and Other Symptoms) of KOOS
Description: as for outcome 1
Time Frame: MACI00206 Baseline and Week 260
Population: Analysis population includes all participants who completed each KOOS subscale at Week 260.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 59
units on a scale
  Change from Baseline Activities of Daily Living | 42.82 [-8.8 to 82.4] | 35.86 [-20.6 to 89.7]
  Change from Baseline Quality of Life | 39.9 [-18.8 to 93.8] | 34.53 [-37.5 to 100]
  Change from Baseline Other Symptoms: number analyzed (Participants) | 65 | 57
  Change from Baseline Other Symptoms | 32.53 [-7.1 to 78.6] | 28.45 [-14.3 to 89.3]

8. Secondary Outcome: Change From MACI00206 Baseline in the Patient's Evaluation of Overall Knee Condition Using the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form
Description: The IKDC Subjective Knee Evaluation Form is a validated knee-specific measure of symptoms, function, and sports activity that is appropriate for patients with a wide variety of knee problems. The form consists of 18 items covering the domains of symptoms, functioning during activities of daily living and sports, and current function of the knee.
  The IKDC Subjective Knee Evaluation Form is scored by summing the scores for the individual items and then transforming the score to a scale that ranges from 0 to 100. The transformed score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
Time Frame: MACI00206 Baseline and Week 260
Population: 64 of the 65 MACI-treated patients and 59 of the 63 microfracture-treated patients enrolled in MACI00809 completed the IKDC form at Week 260.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 64 | 59
units on a scale | 35.48 [-11.5 to 80.5] | 31.58 [-21.8 to 85.1]

9. Secondary Outcome: Change From MACI00206 Baseline in the Patient's Evaluation of Overall Knee Condition Using the Modified Cincinnati Knee Rating System
Description: The Modified Cincinnati Knee Rating System is a self-assessment of the intensity of sports participation, functional limitations, and the ability to participate in different types of sports. The Modified Cincinnati Knee Rating System overall knee condition score ranges from 1 (poor) to 10 (excellent).
Time Frame: MACI00206 Baseline and Week 260
Population: 65 of the 65 MACI-treated patients and 59 of the 63 microfracture-treated patients enrolled in MACI00809 completed the Modified Cincinnati Knee Rating System at Week 260.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 59
units on a scale | 3.55 [-1.0 to 8.0] | 2.71 [-3.0 to 8.0]

10. Secondary Outcome: Change From MACI00206 Baseline in the 12-Item Short-Form Health Survey (SF-12) Physical and Mental Component Scores
Description: The SF-12 is a subset of the 36-Item Short-Form Health Survey (SF-36) and includes 8 subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) that are used to calculate the physical (PCS) and mental (MCS) summary component scores.
  MCS and PCS are summarized as Z-scores using standard SF-12 scoring and a US population means. The Z-score indicates how many standard deviations a score is from the population mean. Higher values reflect better health. Changes from Baseline are reported.
Time Frame: MACI00206 Baseline and Week 260
Population: 65 of the 65 MACI-treated patients and 55 of the 63 microfracture-treated patients enrolled in MACI00809 completed the 12-Item Short-Form Health Survey at Week 260.
Measure: Mean (Full Range); unit: Z-score
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 55
Z-score
  Change from Baseline in Physical Component Score | 1.52 [-1.6 to 4.0] | 1.28 [-1.3 to 3.8]
  Change from Baseline in Mental Component Score | 0.38 [-2.2 to 3.3] | 0.52 [-2.0 to 3.9]

11. Secondary Outcome: Change From MACI00206 Baseline in the European Quality of Life 5 Dimensions (EQ-5D) Visual Analog Scale (VAS) Score
Description: The EQ-5D is a standardized instrument for use as a measure of health outcome (see the EuroQOL Website for details: www.euroqol.org). Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. The EQ Visual Analogue Scale (VAS) was used to record the respondents' self-rated health status on a vertical graduated (0-100) VAS where 0 is 'the worst health you can imagine' and 100 is 'the best health you can imagine'.
Time Frame: MACI00206 Baseline and Week 260
Population: 65 of the 65 MACI-treated patients and 58 of the 63 microfracture-treated patients enrolled in MACI00809 completed the EQ-5D VAS Score at Week 260.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 58
units on a scale | 20.14 [-15.0 to 68.0] | 17.1 [-40.0 to 85.0]

12. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs)
Time Frame: Years 2 through 5 post treatment (MACI or microfracture)
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 63
Participants | 49 | 47

13. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Time Frame: Years 2 through 5 post treatment (MACI or microfracture)
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 63
Participants | 16 | 17

14. Secondary Outcome: Number of Participants Having Subsequent Surgical Procedures (SSPs) in Target Knee
Time Frame: Years 2 through 5 post treatment (MACI or microfracture)
Measure: Count of Participants; unit: Participants
Arm/Group | MACI | Microfracture
Number analyzed (Participants) | 65 | 63
Participants | 7 | 6

ADVERSE EVENTS:
Time Frame: Years 2 through 5 post treatment (MACI or microfracture)
Arm/Group | MACI | Microfracture
Serious Adverse Events (participants affected / at risk) | 16/65 | 17/63
Other Adverse Events (participants affected / at risk) | 49/65 | 46/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MACI (N=65) | Microfracture (N=63)
Cartilage Injury (Injury, poisoning and procedural complications) | 2 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Treatment Failure (General disorders) | 3 | 5 — Adverse events of treatment failure were reported by the Investigator. Not all adverse events of treatment failure met the protocol-specified definition of treatment failure.
Graft delamination (Injury, poisoning and procedural complications) | 1 | 0 — The event of graft delamination was also reported as a treatment failure.
Meniscus Injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Pancreatic injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Ligament laxity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 2
Otosclerosis (Ear and labyrinth disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MACI (N=65) | Microfracture (N=63)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 32
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 5
Joint Effusion (Musculoskeletal and connective tissue disorders) | 2 | 5
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 5
Nasopharyngitis (Infections and infestations) | 7 | 2
Influenza (Infections and infestations) | 4 | 5
Headache (Nervous system disorders) | 11 | 13
Cartilage Injury (Injury, poisoning and procedural complications) | 3 | 5

LIMITATIONS AND CAVEATS:
Potential problems that may be observed with elective participation in extension studies were observed in the SUMMIT Extension. Thus, the value of inferential testing that compares treatment groups without accounting for missing data is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days